CLINICAL TRIAL: NCT01650636
Title: Patient-Partner Stress Management Effects on CFS Symptoms and Neuroimmune Process
Brief Title: Patient-Partner Stress Management Effects on Chronic Fatigue Syndrome Symptoms and Neuroimmune Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael H. Antoni, Principle Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20100771; R01NS072599 (NIH)
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Videophone-delivered stress management intervention; Chronic fatigue syndrome; Symptoms; Neuroimmune processes; Psychosocial
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Stress Management (Experimental)
  Interventions: Behavioral: Patient-Partner Videotelephone-delivered Cognitive Behavioral Stress Management intervention (PP-T-CBSM)
- Health Information (Active Comparator)
  Interventions: Behavioral: Patient-Partner Videotelephone-delivered Health Information (PP-T-HI)

INTERVENTIONS:
Behavioral: Patient-Partner Videotelephone-delivered Health Information (PP-T-HI) — Ten (10) 90-min sessions of Health Information delivered via videophones
  Arms: Health Information
Behavioral: Patient-Partner Videotelephone-delivered Cognitive Behavioral Stress Management intervention (PP-T-CBSM) — Ten (10) 90-min sessions of T-PP-CBSM
  Arms: Cognitive Behavioral Stress Management

SUMMARY:
The purpose of this study is to test the effects of a videotelephone-delivered patient-partner dual-focused cognitive behavioral stress management intervention on chronic fatigue syndrome (CFS) symptoms and related psychosocial and neuroimmune processes in patients diagnosed with chronic fatigue syndrome. Study tests the hypothesis that videophone-delivered patient-partner cognitive behavioral stress management (T-PP-CBSM) intervention improves patient CFS symptoms relative to a videophone-delivered patient-partner Health Information (PP-T- HI) condition.

DETAILED DESCRIPTION:
The study tests the effects of a 10-week patient-partner focused videophone-delivered cognitive behavioral stress management intervention (T-PP-CBSM) intervention (relaxation, stress awareness, cognitive restructuring, coping skills training, interpersonal skills training) versus a time-attention-matched 10-week patient-partner based videophone-delivered health information (T-PP-HI) (health behavior education on nutrition, sleep and other factors) in men and women with chronic fatigue syndrome (CFS) and their partners. The study evaluates the effects of T-PP-CBSM vs T-PP-HI on patient CFS symptoms, neuroimmune processes--diurnal cortisol regulation and immune regulation (pro-inflammatory:anti-inflammatory cytokine ratio ([IL-1β + IL-6 + TNF-α]:[IL-13 + IL-10])-and psychosocial functioning at 5 months and 9 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* men and women diagnosed with chronic fatigue syndrome

Exclusion Criteria:

* no partner
* prior psychiatric treatment for serious psychiatric disorder (e.g., psychosis, suicidality)
* co-morbidity or medical treatment affecting the immune system
* lack of fluency in English

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology University of Miami, Coral Gables, Florida, United States

REFERENCES:
- [Derived] Milrad SF, Hall DL, Jutagir DR, Lattie EG, Czaja SJ, Perdomo DM, Ironson G, Doss BD, Mendez A, Fletcher MA, Klimas N, Antoni MH. Relationship satisfaction, communication self-efficacy, and chronic fatigue syndrome-related fatigue. Soc Sci Med. 2019 Sep;237:112392. doi: 10.1016/j.socscimed.2019.112392. Epub 2019 Jul 16. PMID 31377502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronic Fatigue Syndrome (CFS) and their partners were recruited from CFS physicians clinics and community.
Period: Intervention Phase
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0
Period: Washout up to 5 Months
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Started | 150 | 150
Completed | 141 | 132
Not Completed | 9 | 18
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Physician Decision | 2 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 8
Period: 5 Month Visit
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Started | 141 | 132
Completed | 141 | 132
Not Completed | 0 | 0
Period: Washout up to 9 Months
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Started | 141 | 132
Completed | 135 | 129
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Period: 9 Month Visit
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Started | 135 | 129
Completed | 135 | 129
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Stress Management | Health Information | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 140 | 278
  >=65 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 80 | 158
  Male | 72 | 70 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 49 | 86
  Not Hispanic or Latino | 113 | 101 | 214
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 148 | 146 | 294
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes in Frequency and Severity of CDC-based CFS Symptoms
Description: Changes in the average frequency and average severity ratings of CFS symptoms as assessed by the CDC Symptom Inventory. Participants rated the frequency (1: A little of the time to 5: All of the time) and severity (1: Very mild to 5: Very severe) of individual CFS symptoms. Greater units on the scale indicate greater symptom frequency or severity. The outcome measure was calculated as a set of two composite scores: 1) Average Symptom Frequency, reflecting an aggregated average of frequency across all symptoms, and 2) Average Symptom Severity, reflecting an aggregated average of severity across all symptoms. Change scores are expressed and calculated as Follow-Up minus Baseline scores for average symptom frequency and average symptom severity.
Time Frame: baseline and 5 and 9 month post-intervention follow-up
Population: CFS Patients only were analyzed. (Partner data was not analyzed for this measurement)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
Units on a scale
  Average Symptom Frequency Change at 5 months F/U | 0.29 (0.77) | 0.12 (0.55)
  Average Symptom Frequency Change at 9 months F/U | 0.49 (0.80) | 0.05 (0.67)
  Average Symptom Severity Change at 5 months F/U | 0.46 (0.76) | 0.41 (0.53)
  Average Symptom Severity Change at 9 months F/U | 0.59 (0.80) | 0.34 (0.67)

2. Primary Outcome: Changes in a Single Composite Product of Average Frequency and Severity Scores of CDC-based CFS Symptoms
Description: Changes in the composite product of average frequency and severity scores of CDC-based CFS symptoms assessed by the CDC Symptom Inventory. Participants rated the frequency (1: A little of the time to 5: All of the time) and severity (1: Very mild to 5: Very severe) of individual CFS symptoms. Greater units on the scale indicate greater symptom frequency or severity. The composite outcome measure was calculated as the product of Average Symptom Frequency and Average Symptom Severity. Change scores are expressed and calculated as Follow-Up minus Baseline scores for the composite product score.
Time Frame: baseline and 5 and 9 months post-intervention follow-up
Population: CFS Patients only were analyzed. (Partner data was not analyzed for this measurement)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
Units on a scale
  (Frequency * Severity) Change at 5 months F/U | 1.65 (3.37) | 1.37 (2.38)
  (Frequency * Severity) Change at 9 months F/U | 2.62 (3.87) | 1.10 (3.31)

3. Secondary Outcome: Changes in Neuroimmune Functioning Measured by Change in Averaged (2-day) Di-urnal Slope of Salivary Cortisol.
Description: Changes in salivary cortisol diurnal pattern is measured to determine changes in neuroimmune function. Salivary cortisol diurnal pattern is computed as the natural log of the average within-day slope of change over the 2-day collection period. This measurement is made at baseline, 5 month follow-up and 9 month follow-up. Outcomes are expressed as change in Cortisol Diurnal Pattern (natural log of average 2-day slope values) and expressed and calculated as Follow-Up minus Baseline values (using the natural log of average 2-day slope values).
Time Frame: baseline and 5 and 9 month post-intervention follow-up
Population: CFS Patients only were analyzed. (Partner data was not analyzed for this measurement)
Measure: Mean (Standard Deviation); unit: Ug/dL
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
Ug/dL
  Change at 5 months F/U | 0.24 (1.19) | -0.06 (1.25)
  Change at 9 months F/U | 0.08 (1.19) | 0.31 (1.86)

4. Secondary Outcome: Changes in Neuroimmune Functioning Measured by Pro-Inflammatory Cytokines
Description: Serum samples were collected to measure the pro-inflammatory cytokines Interleukin (IL)-1a, IL-6 and Tumor Necrosis Factor (TNF)-a for neuroimmune function. Units of measure are raw concentration expressed picograms per milliliter (pg/mL). Change values are expressed and calculated as Follow-Up minus Baseline values (using raw values).
Time Frame: Baseline, 5 months, 9 months
Population: CFS Patients Only were analyzed. Data for this outcome measure were not collected from partners.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
pg/mL
  IL-1a Change at 5 months F/U | 0.39 (8.25) | 0.10 (8.33)
  IL-1a Change at 9 months F/U | 0.42 (6.68) | -0.32 (7.27)
  IL-6 Change at 5 months F/U | 0.84 (6.88) | -0.59 (5.09)
  IL-6 Change at 9 months F/U | 0.43 (3.61) | -0.30 (5.36)
  TNFa Change at 5 months F/U | -1.34 (15.86) | 4.28 (19.64)
  TNFa Change at 9 months F/U | -2.52 (14.86) | -1.05 (22.87)

5. Secondary Outcome: Changes in Neuroimmune Functioning Measured by Anti-inflammatory Cytokines
Description: Serum samples were collected to measure the anti-inflammatory cytokines Interleukin (IL)-4, IL-5 and IL-10 for neuroimmune function. Units of measure are raw concentration expressed picograms per milliliter (pg/mL). Change values are expressed and calculated as Follow-Up minus Baseline values (using raw values).
Time Frame: Baseline, 5 months, 9 months
Population: Only CFS Patients were analyzed. Partner data was not collected for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
pg/mL
  IL-4 Change at 5 months F/U | 0.61 (3.93) | 0.54 (3.03)
  IL-4 Change at 9 months F/U | -0.06 (3.09) | 0.37 (2.27)
  IL-5 Change at 5 months F/U | -0.42 (3.26) | -0.23 (4.28)
  IL-5 Change at 9 months F/U | -1.05 (4.73) | -0.55 (3.99)
  IL-10 Change at 5 months F/U | -1.02 (10.53) | -0.77 (10.30)
  IL-10 Change at 9 months F/U | 1.01 (10.90) | 2.67 (26.26)

6. Secondary Outcome: Changes in Neuroimmune Regulation Measured by Ratio of Pro-Inflammatory to Anti-Inflammatory Cytokines
Description: Serum samples were collected to measure the pro-inflammatory:anti-inflammatory cytokine ratio ([IL-1β + IL-6 + TNF-α]:[IL-13 + IL-10]) for neuroimmune function. These values are expressed as ratios. Change values are expressed and calculated as Follow-Up minus Baseline values (using ratio values).
Time Frame: baseline and 5 and 9 months post-intervention follow-up
Population: CFS Patients only were analyzed. (Partner data was not analyzed for this measurement)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
Ratio
  Ratio Change at 5 months F/U | -0.43 (5.28) | -0.38 (8.55)
  Ratio Change at 9 months F/U | 0.23 (6.98) | -1.14 (13.73)

7. Secondary Outcome: Changes in Psychosocial Functioning
Description: Changes in psychosocial functioning measured with the Perceived Stress Scale (PSS), Center for Epidemiologic Studies-Depression (CES-D) scale, and the subscales of the Sickness Impact Profile (SIP) for Recreation and Pastimes, and Social Interaction. Greater scores on the PSS indicate greater perceived stress (range: 0-56) and greater scores on the CES-D indicate greater depressive symptoms (range: 0-60). The SIP is divided into 'Social Interaction' and 'Recreation and Pastimes' subscales (ranges: 0-11 and 0-5, respectively), with greater scores indicating greater impact of sickness in the respective domain. Change scores are expressed and calculated as Follow-Up minus Baseline scores.
Time Frame: baseline and 5 and 9 month post-intervention follow-up
Population: Only CFS Patient's data were analyzed. Partner data was not collected for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cognitive Behavioral Stress Management | Health Information
Number analyzed (Participants) | 75 | 75
Units on a scale
  PSS Change at 5 months F/U | -2.57 (8.17) | -2.84 (7.39)
  PSS Change at 9 months F/U | -0.56 (9.07) | -3.28 (8.30)
  CES-D Change at 5 months F/U | -0.44 (10.67) | -1.36 (10.18)
  CES-D Change at 9 months F/U | 1.66 (12.20) | -3.08 (11.21)
  SIP Recreation and Pastimes Change at 5 months F/U | -0.95 (3.78) | -0.98 (2.80)
  SIP Recreation and Pastimes Change at 9 months F/U | -0.23 (3.32) | -0.70 (3.50)
  SIP Social Interaction Change at 5 months F/U | 0.95 (3.78) | 0.98 (2.80)
  SIP Social Interaction Change at 9 months F/U | 0.23 (3.32) | 0.70 (3.50)

ADVERSE EVENTS:
Time Frame: Adverse event collected for the duration of the study and up to 9 months.
Arm/Group | Cognitive Behavioral Stress Management | Health Information
All-Cause Mortality (participants affected / at risk) | 1/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 1/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 2/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Stress Management (N=150) | Health Information (N=150)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Stress Management (N=150) | Health Information (N=150)
Rotator Cuff Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT01650636/Prot_SAP_000.pdf